CLINICAL TRIAL: NCT06478706
Title: A Randomised, Double-Blind, Placebo Controlled, Two-Part Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of a Repeat Dose of Inhaled ETD001 in People With Cystic Fibrosis
Brief Title: A Two-Part Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Repeat Doses of Inhaled ETD001 in People With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enterprise Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-ENAC-03
Record Dates: First submitted 2024-06-18; First posted 2024-06-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A - 7 day treatment period - parallel group (Experimental): Twice daily doses of ETD001/placebo for 6 days, single dose on Day 7
  Interventions: Drug: ETD001; Drug: Placebo
- Part B - 2 x 28 day treatment period - crossover (Experimental): Two treatment periods of twice daily doses of ETD001/placebo for 27 days, single dose on Day 28 separated by a period of 28 days
  Interventions: Drug: ETD001; Drug: Placebo

INTERVENTIONS:
Drug: ETD001 — Twice daily doses
Drug: Placebo — Twice daily doses

SUMMARY:
This study is the first to give ETD001 to people with CF. The study will be run in two parts. Part A will assess if ETD001 is safe to give to people with CF, and Part B will assess if ETD001 improves lung function. The study drug is taken twice a day, in Part A it is taken for 7 days and in Part B for 28 days. In Part B there will be a separate period where dummy medicine is given for 28 days so the treatments can be compared.

In Part A participants will receive 13 doses of either ETD001 or placebo, 8 people will take part. Participants will take up to 56 days to finish the study and make 5 outpatient visits.

In Part B participants will receive 55 doses of ETD001 and 55 doses of placebo, 32 people will take part. Participants will take up to 140 days to finish the study and will make 8 outpatient visits.

Study assessments include physical examinations, vital signs, heart traces, blood/urine samples, breathing tests and health questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male & female ≥ 18 years of age, who fit one of the following criteria:

Women of childbearing potential using permitted contraception a minimum of 28 days before dosing until completion of the final follow up visit; Women of non-childbearing potential; Men using contraception from the time of the first dose, until completion of the final follow up visit;

* Confirmed diagnosis of CF
* FEV1 ≥ 40% and ≤ 90% of predicted normal for age, gender, and height
* Able to reproducibly perform spirometry manoeuvres
* Clinically stable CF lung disease
* Routine CF therapy has not changed within 28 days prior to screening.
* Provided written informed consent.
* Body mass index (BMI) > 16 and < 30 kg/m2

Exclusion Criteria:

* Abnormal liver function
* Abnormal renal function
* History of solid organ transplant
* Chest x-ray within the past 12 months with abnormalities suggesting unstable pulmonary disease other than CF
* Received CFTR modulator therapy in the 60 days before screening
* Changes in bronchodilator, corticosteroid or other anti-inflammatory medications 14 days before screening
* Unable to withhold use of long-acting bronchodilators 24 hours or short-acting bronchodilators 6 hours before spirometry assessments
* Unable to withhold use of anti-cholinergics within 24 hours of spirometry
* Started dornase alfa, hypertonic saline, or other airway clearing therapy less than 28 days before screening
* Using inhaled antibiotics for less than 2 complete cycles and unable to complete the entire study during the off or on cycle.
* Changes in inhaled or oral antibiotic use within 14 days of screening
* Taking oral corticosteroids in excess of 10 mg/day or 20 mg every other day within 14 days of screening
* Use of diuretics, or renin-angiotensin aldosterone system antihypertensive drugs , drospirenone, or trimethoprim in the 28 days before screening
* Presence of co-morbidities and medical history in the opinion of the investigator, may pose additional risk by participating in the study, or may confound the results of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and tolerability of repeat inhaled doses of ETD001 monitored by assessment of adverse events | 28 days
  Incidence of treatment emergent adverse events(AE)/serious AE), withdrawals due to AE
Part B: Effect of repeat inhaled doses of ETD001 on percent predicted forced expiratory volume in 1 second (ppFEV1) | Treatment Period 1 & 2 - Day 1 (pre-dose, 1, 2 & 4 hours post dose), Day 14 (pre-dose, 1 & 2 hours post), Day 28 (at 0, 1, 2 & 4 hours post dose)
  Change in ppFEV1 measured by spirometry from baseline to Day 28 (for either Treatment Period 1 or Treatment Period 2), compared to placebo

SECONDARY OUTCOMES:
Part A: Characterisation of plasma pharmacokinetics (PK) | Day 1 (pre-dose, 0.25, 0.5, 1, 2, 4 & 6 hours)
  Peak plasma concentration and time observed (Cmax & Tmax) of ETD001 following dosing.
Part A: Characterisation of plasma pharmacokinetics (PK) | Day 1 (pre-dose, 0.25, 0.5, 1, 2, 4 & 6 hours, Day 7 (pre-dose), Day 28 (single sample)
  Area under the concentration versus time curve from time 0 to last quantifiable concentration (AUC(0-t)) of ETD001 following dosing.
Part A: Characterisation of plasma pharmacokinetics (PK) | Day 1 (pre-dose, 0.25, 0.5, 1, 2, 4 & 6 hours, Day 7 (pre-dose)
  Area under the concentration versus time curve within a dosing interval (AUC(0-tau)) of ETD001 following dosing.
Part A: Characterisation of plasma pharmacokinetics (PK) | Day 1 (pre-dose, 0.25, 0.5, 1, 2, 4 & 6 hours, Day 7 (pre-dose) Day 28 (single sample)
  Area under the concentration versus time curve from time 0 to infinity (AUC(inf)) of ETD001 following dosing.
Part A: Characterisation of plasma pharmacokinetics (PK) | Day 1 (pre-dose, 0.25, 0.5, 1, 2, 4 & 6 hours, Day 7 (pre-dose), Day 28 (single sample)
  Apparent terminal rate constant and apparent terminal half life (λz, T1/2) of ETD001 following dosing.
Part A: Characterisation of urine PK | Day 1 (0 - 6 hours)
  Amount ETD001 excreted in urine (Ae)
Part A: Characterisation of urine PK | Day 1 (0 - 6 hours)
  Fraction of ETD001 dose excreted (Fe)
Part A: Characterisation of urine PK | Day 1 (0 - 6 hours)
  Renal clearance of ETD001 (CLr)
Part B: Effect of repeat inhaled doses of ETD001 on other lung function assessments | Treatment Period 1 & 2; Day 1 (pre-dose, 1, 2 & 4 hours), Day 14 (pre-dose, 1 & 2 hours), Day 28 (pre-dose, 1, 2 & 4 hours)
  Relative change in ppFEV1, absolute change in FVC, FEV1/FVC ratio and FEF25-75 measured by spirometry, from baseline to Day 28 (for either Treatment Period 1 or Treatment Period 2), compared to placebo
Part B: Safety and tolerability of repeat inhaled doses of ETD001 monitored by assessment of adverse events | 105 days
  Incidence of treatment emergent adverse events(AE)/serious AE), withdrawals due to AE
Part B: Effect of repeat inhaled doses of ETD001 on the quality of life questionnaire, the Cystic Fibrosis Questionnaire (revised) (CFQ-R) | Treatment Period 1 & 2; Day 1 & Day 28 (pre-dose)
  Change in CFQ-R (respiratory domain) from baseline to Day 28 (for either Treatment Period 1 or Treatment Period 2), compared to placebo
Part B: Characterisation of plasma PK | Treatment Period 1 & 2; Day 1 (0 & 1 hour), Day 14 (0 & 2 hours), Day 28 (0 & 4 hours), Follow up (Day 105) 1 sample
  Population PK characteristics and model generated individual PK parameters (Cmax & Tmax)
Part B: Characterisation of plasma PK | Treatment Period 1 & 2; Day 1 (0 & 1 hour), Day 14 (0 & 2 hours), Day 28 (0 & 4 hours), Follow up (Day 105) 1 sample
  Population PK characteristics and model generated individual PK parameters (AUC(0-t))
Part B: Characterisation of plasma PK | Treatment Period 1 & 2; Day 1 (0 & 1 hour), Day 14 (0 & 2 hours), Day 28 (0 & 4 hours), Follow up (Day 105) 1 sample
  Population PK characteristics and model generated individual PK parameters (AUC(0-tau))
Part B: Characterisation of plasma PK | Treatment Period 1 & 2; Day 1 (0 & 1 hour), Day 14 (0 & 2 hours), Day 28 (0 & 4 hours), Follow up (Day 105) 1 sample
  Population PK characteristics and model generated individual PK parameters (AUC(0-inf))
Part B: Characterisation of plasma PK | Treatment Period 1 & 2; Day 1 (0 & 1 hour), Day 14 (0 & 2 hours), Day 28 (0 & 4 hours), Follow up (Day 105) 1 sample
  Population PK characteristics and model generated individual PK parameters (λz, T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Renu Gupta, MD, Study Director — Enterprise Therapeutics
Locations (21):
- France (4):
  - Hospices Civils de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - Hôpital Cochin, Paris
  - Hôpitaux de Toulouse, Toulouse
- Germany (6):
  - Charité Universtaetsmedizin, Berlin
  - CF-Studienzentrum Universitätsklinikum Köln, Cologne
  - Westdeutsches Lungenzentrum am Universitätsklinikum, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - IKF Pneumologie, Frankfurt
  - LMU Kinikum, Munich
- Italy (5):
  - Azienda Ospedaliera Universitaria Meyer, Florence
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda- Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- United Kingdom (6):
  - Belfast Health and Social Care Trust, Belfast
  - Royal Papworth Hospital, Cambridge
  - All Wales Adult CF Centre, Cardiff
  - Queen Elizabeth University Hospital West of Scotland CF Service, Glasgow
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton